CLINICAL TRIAL: NCT05712850
Title: A Prospective, Single Arm Clinical Trial Evaluating Clinical Outcome and Fusion Results Using the SiJoin® Transfixing Sacroiliac Fusion Device
Brief Title: Clinical Outcome and Fusion Results Using the SiJoin® Transfixing Sacroiliac Fusion Device
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: VG Innovations, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: VGI-004
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Sacroiliitis; Sacroiliac Joint Dysfunction; Iatrogenic Injury; Osteitis Condensans Ilii; Pelvic Fracture
MeSH Terms: conditions — Sacroiliitis; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: SiJoin® Transfixing Sacroiliac Fusion Device — Sacroiliac Fusion

SUMMARY:
The purpose of this clinical study is to evaluate fusion of the SI joint(s) and any reduction in VAS pain scores in a prospective cohort of patients utilizing the SiJoin® Transfixing Sacroiliac Fusion Device in patients that received sacroiliac fusion, without ancillary stabilization devices.

DETAILED DESCRIPTION:
Study Title: A prospective, single arm clinical trial evaluating clinical outcome and fusion results using the SiJoin® Transfixing Sacroiliac Fusion Device

Instrumentation SiJoin® Transfixing Sacroiliac Fusion Device Study Design: Non-randomized, prospective, single arm, single center clinical trial

Patient Population and Sample Size:

Patients (n≥25) from 1 clinical site, who have been medically evaluated, found appropriate for, and have agreed to treatment by sacroiliac joint fixation, including unilateral and/or bilateral sacroiliac fusion according to accepted medical standards using the SiJoin® Transfixing Sacroiliac Fusion Device.

Objectives: The primary objective of this study is:

1. Evaluate the fusion status of sacroiliac joints at 12 months (depending on patient (vailability) following joint fusion/fixation using the SiJoin® Transfixing Sacroiliac Fusion Device;
2. Subject success / Clinical outcome: Evaluate the reduction in baseline VAS back pain score at 2-3 weeks, 3 months, and 12 months.

The secondary objectives of this study are to:

1. Assess the ease of use of the SiJoin® Fusion System;
2. Document the occurrence of adverse events related or possibly related to the use of the SiJoin® Fusion System;
3. Document the occurrence of subsequent surgical intervention at the sacroiliac joint.

Inclusion Criteria:

Candidates must meet ALL of the following:

1. Have provided consent for research by signing the Information and Consent for Research form;
2. Have given appropriate operative consent for a sacroiliac joint fixation procedure as standard of care using the SiJoin® Transfixing Sacroiliac Fusion Device;
3. Are skeletally mature male or female, and are at least 18 years of age at time of surgery;
4. Patient history confirms sacroiliac joint disfunction;
5. Failure of six months of conservative care;
6. Failure of NSAIDs;
7. Positive diagnosis injection of sacroiliac joint; and
8. Agree to adhere to post-surgical medically prescribed activity limitations and/or physical rehabilitation.

Exclusion Criteria:

Candidates will be excluded if they have ANY of the following:

1. Previous surgery or prior hardware in place at the target sacroiliac joint;
2. Deidentified data cannot be provided;
3. If female, pregnant at time of sacroiliac joint surgery;
4. Found to be inappropriate candidate for sacroiliac joint fixation;
5. Requires additional and/or other surgical technique and/or approach to the sacroiliac joint, which may in the opinion of the Primary Investigator confound measurement of outcome variables;
6. Has a medical disorder or is receiving medications that would be expected to interfere with osteogenesis;
7. Has active malignancy, or patient with a history of any malignancy (except non-melanoma skin cancer) with recurrence within 5 years or surgery;
8. Has active local or systemic infection or history of local or systemic infection, immune-deficiency, uncontrolled medical conditions, which in the opinion of the Investigator may increase patient risk or confound fusion results;
9. Has BMI >40%;
10. Has history of tobacco smoking within 6 months prior to operation;
11. Has history of alcoholism, medication or drug abuse, psychosis, is a prisoner, and/or has a personality disorder, poor motivation, emotional or intellectual issues that would likely make the patient unreliable for participation in the study;
12. Has history of diabetes;
13. Are participating in any other clinical trial;
14. Patient is an employee (or family members of employees) of the PI/site or Sponsor; or
15. Patient is limited or non-reader (e.g., blind, illiterate) Study Duration: 12 months

Study Outcomes:

The primary study outcomes of this study are:

1. Fusion grade at 12 months follow-up (depending on patient availability) using CT scans with a grading system based on:

   1. Complete fusion; or
   2. No fusion.
2. Subject success / Clinical outcome: Evaluate the reduction in baseline VAS back pain score at:

   1. 2-3 weeks;
   2. 3 months; and
   3. 12 months.

The secondary outcomes of this study are:

1. Surgeon opinion of "ease of use" utilizing the SiJoin® Fusion System;
2. Occurrence of adverse events related or possibly related to the use of the SiJoin® Fusion System; and
3. Occurrence of subsequent surgical intervention at the target joint.

Study Assessments

* Intraoperative: Post-placement radiograph;
* 12 month: sacroiliac joint CT scan;
* Patient provided VAS pain scores at pre-op, and each subsequent follow-up appointment.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided consent for research by signing the Information and Consent for research form;
2. Have given appropriate operative consent for a sacroiliac joint fixation procedure as standard of care using the SiJoin® Transfixing Sacroiliac Fusion Device;
3. Are skeletally mature male or female, and are at least 18 years of age at time of surgery;
4. Patient history confirms sacroiliac joint disfunction;
5. Failure of six months of conservative care;
6. Failure of NSAIDs;
7. Positive diagnosis injection of sacroiliac joint; and
8. Agree to adhere to post-surgical medically prescribed activity limitations and/or physical rehabilitation.

Exclusion Criteria:

1. Previous surgery or prior hardware in place at the target sacroiliac joint;
2. Deidentified data cannot be provided;
3. If female, pregnant at time of sacroiliac joint surgery;
4. Found to be inappropriate candidate for sacroiliac joint fixation;
5. Requires additional and/or other surgical technique and/or approach to the sacroiliac joint, which may in the opinion of the Primary Investigator confound measurement of outcome variables;
6. Has a medical disorder or is receiving medications that would be expected to interfere with osteogenesis;
7. Has active malignancy, or patient with a history of any malignancy (except non-melanoma skin cancer) with recurrence within 5 years or surgery;
8. Has active local or systemic infection or history of local or systemic infection, immune-deficiency, uncontrolled medical conditions, which in the opinion of the Investigator may increase patient risk or confound fusion results;
9. Has BMI >40%;
10. Has history of tobacco smoking within 6 months prior to operation;
11. Has history of alcoholism, medication or drug abuse, psychosis, is a prisoner, and/or has a personality disorder, poor motivation, emotional or intellectual issues that would likely make the patient unreliable for participation in the study;
12. Has history of diabetes;
13. Are participating in any other clinical trial;
14. Patient is an employee (or family members of employees) of the PI/site or Sponsor; or
15. Patient is limited or non-reader (e.g., blind, illiterate)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been evaluated and found appropriate for SI joint fixation according to accepted medical standards, and have agreed to this surgical procedure will be considered for study enrollment. Only those patients judged by the surgeon (intra-operatively) to be suitable for SI joint fixation using the SiJoin® Transfixing Sacroiliac Fusion Device will be included in data collection.
  Study patients will be identified and recruited from outpatient facilities affiliated with investigative sites. For the purposes of enrollment, patients will only be considered evaluable study patients after they complete eligibility screening and sign the study Information and Consent for Research Form.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-01-18 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Fusion Status/Evaluation | 12 Months
  Evaluate the fusion status of SI Joints using CT scans with a grading system based on:
  1. Complete fusion; or
  2. No fusion.
Visual Analog Scale (VAS) Reduction | 2-3 weeks, 3 Months, 6 Months, 12 Months
  Scale: 0 (No Pain) - 10 (Worst Pain Possible)
  Composite endpoint of reduction from baseline in VAS back pain score by at least 2 points.

SECONDARY OUTCOMES:
Ease of Use | 12 months
  Assess the ease of use of the SiJoin® Fusion System
  Scale: 0 (Easy) - 10 (Extremely Difficult)
Adverse Avents | 12 months
  Monitor the occurrence of adverse events related or possibly related to the use of the SiJoin® Fusion System;
Subsequent Surgical Interventions | 12 months
  Monitor the occurrence of subsequent surgical intervention at the target sacroiliac joint(s).

CONTACTS AND LOCATIONS:
Locations (1):
- Seaside Surgery Center, Naples, Florida, United States